CLINICAL TRIAL: NCT05088707
Title: Sublingual Versus Vaginal Misoprostol In Medical Treatment of Second Trimestric Missed Miscarriage: A Randomized Controlled Trial
Brief Title: Sublingual Versus Vaginal Misoprostol In Medical Treatment of Second Trimestric Missed Miscarriage
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Aswan University Hospital (Other)
Responsible Party: Principal Investigator, hany farouk, A Professor, Aswan University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: aswu/354/3/18
Record Dates: First submitted 2021-10-10; First posted 2021-10-22 (Actual); Last update posted 2021-10-22 (Actual); Status verified 2021-10

CONDITIONS: Miscarriage
Keywords: miscarriage; sublingual; vaginal; misoprostol
MeSH Terms: conditions — Abortion, Spontaneous

STUDY DESIGN:
Intervention Model Description: an open-label randomized controlled study
Masking Description: an open-label randomized controlled study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sublingual misoprostol (Experimental): All patients will receive three doses of sublingual misoprostol every four hours. The first dose of misoprostol 800 mcg will be administrated at the hospital. Then the patient will be observed for 1 hour for any immediate adverse reaction Clear instructions about the method and timing of the second dose will be given upon sending home.
  Two doses of misoprostol 800 mcg each (four tablets of 200 mcg per dose). Paracetamol, eight hourly, will be provided as an analgesic or antipyretic. A specimen bottle to collect the POC if passed out. Two pairs of disposable gloves. Pre-filled histopathological examination form to be sent to the laboratory together with the products of conception
  Interventions: Drug: sublingual misoprostol
- vaginal misoprostol (Active Comparator): All patients will receive three doses of vaginal misoprostol every four hours The first dose of misoprostol 800 mcg will be administrated at the hospital. Then the patient will be observed for 1 hour for any immediate adverse reaction Clear instructions about the method and timing of the second dose will be given upon sending home.
  Paracetamol, eight hourly, will be provided as analgesic or antipyretic
  Interventions: Drug: vaginal misoprostol

INTERVENTIONS:
Drug: sublingual misoprostol — All patients will receive three doses of sublingual misoprostol every four hours The first dose of misoprostol 800 mcg will be administrated at the hospital. Then the patient will be observed for 1 hour for any immediate adverse reaction Clear instructions about the method and timing of second dose will be given upon sending home.
  Two doses of misoprostol 800 mcg each (four tablets of 200 mcg per dose). Paracetamol, eight hourly, will be provided as analgesic or antipyretic. A specimen bottle to collect the POC if passed out. Two pairs of disposable gloves. Pre-filled histopathological examination form to be sent to the laboratory together with the products of conception
  Other Names: experimental
  Arms: sublingual misoprostol
Drug: vaginal misoprostol — All patients will receive three doses of vaginal misoprostol every four hours The first dose of misoprostol 800 mcg will be administrated at the hospital. Then the patient will be observed for 1 hour for any immediate adverse reaction Clear instructions about the method and timing of the second dose will be given upon sending home.
  Paracetamol, eight hourly, will be provided as analgesic or antipyretic
  Other Names: Active Comparator
  Arms: vaginal misoprostol

SUMMARY:
The aim of this work is to compare the effectiveness of vaginal versus sub-lingual misoprostol for medical treatment of the second trimester missed miscarriage

DETAILED DESCRIPTION:
In women with second trimester-missed miscarriage, sublingual misoprostol may be as vaginal misoprostol in the achievement of successful miscarriage so our aim was to compare the effectiveness of vaginal versus sub-lingual misoprostol for medical treatment of the second trimester missed miscarriage.

ELIGIBILITY:
Inclusion Criteria:

* All women above 18 years of age
* between 13-26 weeks of gestation.
* Pregnancy is confirmed by a pregnancy test or ultrasound scan.
* missed abortion
* Normal general and gynecological examination.

Exclusion Criteria:

* Hemodynamically unstable.
* Suspected sepsis with temperature 38 °C.
* Concurrent medical illness e.g. hematological, cardiovascular, thromboembolism,
* respiratory illnesses, recent liver disease, or pruritus of pregnancy.
* Presence of intrauterine contraceptive device (IUCD).
* Suspect or proven ectopic pregnancy.
* -Failed medical or surgical evacuation before the presentation.
* Known allergy to misoprostol.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — pregnant women with second missed abortion
Enrollment: 200 (Estimated)
Dates: Start 2021-11-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Completeness of abortion | 7 days
  expulsion of Products of conception by visual inspection

SECONDARY OUTCOMES:
Successful medical abortion | 7 days
  cervical os is closed with endometrial thickness of less than 15 mm
Bleeding pattern following treatment | 7 days
  This will be assessed by hemoglobin(g/dl) and haematocrit level after the treatment , if the patients required blood transfusion and number of units transfused and number of days of bleeding

CONTACTS AND LOCATIONS:
Locations (1):
- Aswan University Hospital, Aswān, Egypt

IPD SHARING:
Plan to Share IPD: No